CLINICAL TRIAL: NCT03313284
Title: Acute Effects of Intermittent Respiratory Muscle Training and Hypoxia on Cardiovascular and Sleep Parameters in Elderly Persons With Prehypertension
Brief Title: Respiratory Muscle Training and Intermittent Hypoxia: Additive Health Effects?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REHYPE_2017
Record Dates: First submitted 2017-10-04; First posted 2017-10-18 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Pre-Hypertension
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental)
  Interventions: Procedure: RMT; Procedure: RMT + IH; Procedure: Control

INTERVENTIONS:
Procedure: RMT — RMT consists of six bouts of 5-min of volitional hyperpnoea . After each RMT bout, participants will breathe room air for 5 minutes.
Procedure: RMT + IH — RMT and IH consist of six bouts of 5-min of volitional hyperpnoea. After each RMT bout, participants will breathe a hypoxic gas mixture (10.5% O2 ) for 5 minutes.
Procedure: Control — No intervention

SUMMARY:
The prevalence of pre-hypertension and hypertension in the elderly is very high. Apart from medication, physical exercise training is a potential strategy to reduce blood pressure, however, the ability to perform exercise can be limited in the elderly. Hence, alternative non-pharmacological strategies to reduce blood pressure are necessary. Two interventions that have been shown to positively influence blood pressure are respiratory muscle training (RMT) and intermittent hypoxia (IH). Whether a combination of RMT and IH yields even better effects is currently unknown. Therefore, in this study, the effect of a single session of RMT with and without IH on blood pressure and associated cardiovascular parameters will be investigated in elderly subjects with pre-hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age: 65-80 years
* Systolic blood pressure between 130-139 mmHg and diastolic blood pressure lower than 90 mmHg
* Non smoking
* Normal Body-Mass-Index (BMI): 18.5-24.9 kg·m-2
* Normal Lung Function
* Willing to adhere to the general study rules

Exclusion Criteria:

* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Intake of blood pressure medication
* Intake of medications affecting sleep or the performance or the respiratory, cardiovascular or neuromuscular system
* Acute or chronic illness other than prehypertension

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure in mmHg | At baseline after 20 min of lying in a supine position, every 5 minutes during the 60 min intervention, and 20, 35 and 50 min after the end of the intervention
  Blood pressure before, during, and after each intervention measured with an automated sphygmomanometer

SECONDARY OUTCOMES:
Change in pulse wave velocity in m/s | At baseline after 25 min of lying in a supine position, and 25, 40 and 55 min after the end of the intervention
  Carotid-femoral pulse wave velocity before and after each intervention, assessed with a device that simultaneously records (non-invasively) pressure signals from the carotid and femoral arteries
Change in cardiac output in L/min | At baseline after 15min of lying in a supine position, every 5 minutes during the 60 min intervention, and 15, 30 and 45 min after the end of the intervention
  Cardiac output before, during, and after each intervention measured with impedance cardiography
Change in total peripheral resistance in dyn x s/cm^5 | At baseline after 15min of lying in a supine position, every 5 minutes during the 60 min intervention, and 15, 30 and 45 min after the end of the intervention
  Total peripheral resistance before, during, and after each intervention measured with impedance cardiography
Changes in baroreflex sensitivity in ms/mmHg | At baseline after 15min of lying in a supine position, and 15, 30 and 45 min after the end of the intervention
  Baroreflex sensitivity before and after each intervention assessed with photo plethysmography
Change in heart rate variability in ms | At baseline after 15min of lying in a supine position, every 5 minutes during the 60 min intervention, and 15, 30 and 45 min after the end of the intervention
  Heart rate variability measured before, during and after each intervention with impedance cardiography
Change in peripheral oxygenation during sleep in %Saturation | Continuously during the night following each intervention, from time to bed until wake up time in the morning (i.e. on average approximately 8hours)
  Peripheral oxygenation during sleep measured at home after each intervention with a finger pulse oxymeter
Change in sleep efficiency defined as the ratio of total sleep time and time in bed | Continuously during the night following each intervention, from time to bed until wake up time in the morning (i.e. on average approximately 8hours)
  Sleep efficiency measured at home after each intervention with an actigraph
Change in subjective sleep quality | Within 5 minutes after waking-up following the night after each intervention
  Sleep quality (i.e. "How well did you sleep?" and "How recovered are you?") measured at home after each intervention with a visual analog scale (VAS). The two VAS consists each of a 10cm-horizontal line, with the left end of the lines representing low sleep quality ("slept very badly" and "not recovered at all", respectively) and the right end representing good sleep quality ("slept very well" and "completely recovered", respectively). Participants are asked to draw a vertical line in between the two ends on each of the two VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Christina M. Spengler, Prof., Principal Investigator — Exercise Physiology Lab, Institute of Human Movement Sciences and Sport, ETH Zurich
Locations (1):
- Exercise Physiology Lab, Institute of Human Movement Sciences and Sport, ETH Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No